CLINICAL TRIAL: NCT01213836
Title: A Phase IV Prospective, Double-blind, Double-dummy, Randomised, Crossover Study to Assess the Impact on Daily Cognitive Functioning of Quetiapine Fumarate Immediate Release (Seroquel IR®) Dosed Twice Daily and Quetiapine Fumarate Extended Release (Seroquel XR®) Dosed Once Daily in the Evening in Patients With Stable Schizophrenia
Brief Title: Compare the Effect on Cognitive Functioning of Two Formulations of Seroquel, Seroquel XR and IR in Patients With Stable Schizophrenia
Acronym: eXtRa
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: D1443L00082; 2010-020579-21 (EudraCT Number)
Record Dates: First submitted 2010-10-01; First posted 2010-10-04 (Estimated); Results first posted 2012-07-27 (Estimated); Last update posted 2012-07-27 (Estimated); Status verified 2012-05

CONDITIONS: Schizophrenia
Keywords: Stable schizophrenia; cognitive functioning
MeSH Terms: conditions — Schizophrenia

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- First Seroquel XR then Seroquel IR (Active Comparator): Patients randomised to Seroquel XR will have treatment for 10-16 days and after that cross-over to treatment with Seroquel IR for 10-16 days
  Interventions: Drug: Seroquel XR- quetiapine fumarate extended release; Drug: Seroquel IR - quetiapine fumarate; Drug: Placebo matching Seroquel XR; Drug: Placebo matching Seroquel IR
- First Seroquel IR then Seroquel XR (Active Comparator): Patients randomised to Seroquel IR will have treatment for 10-16 days and after that cross-over to treatment with Seroquel XR for 10-16 days
  Interventions: Drug: Seroquel XR- quetiapine fumarate extended release; Drug: Seroquel IR - quetiapine fumarate; Drug: Placebo matching Seroquel XR; Drug: Placebo matching Seroquel IR

INTERVENTIONS:
Drug: Seroquel XR- quetiapine fumarate extended release — Seroquel XR dose 400-700 mg (in tablet form). The investigator established the dosing schedule for each patient depending on the patient's dose when entering the study. The patients continued on the same dose during the study as they had prior to enrolment. Dose taken once a day for 10-16 days.
Drug: Seroquel IR - quetiapine fumarate — Seroquel IR dose 400-700 mg (in tablet form). The investigator established the dosing schedule for each patient depending on the patient's dose when entering the study. The patients continued on the same dose during the study as they had prior to enrolment. Dose taken twice a day for 10-16 days.
Drug: Placebo matching Seroquel XR — Placebo matching Seroquel XR dose 400-700 mg (in tablet form). Dose taken once a day for 10-16 days.
Drug: Placebo matching Seroquel IR — Placebo matching Seroquel IR dose 400-700 mg (in tablet form). Dose taken twice a day for 10-16 days.

SUMMARY:
This will be a phase IV 20 -32 day prospective, double blind, double-dummy, randomised crossover study that will evaluate the effect of quetiapine XR and quetiapine IR on cognitive performance in patients with schizophrenia stabilized on a single antipsychotic medication.

ELIGIBILITY:
Inclusion Criteria:

* Provision of written informed consent prior to any study specific procedures
* Documented clinical diagnosis of schizophrenia, paranoid type, for at least 2 years before randomisation meeting the Diagnostic and Statistical Manual of Mental Disorders, 4th Edition (DSM-IV, American Psychiatric Association 2000) criteria of schizophrenia (DSM-IV codes 295.3) confirmed by MINI version 5.0
* Outpatient status at enrolment
* Dose of quetiapine IR or quetiapine XR unchanged during the last 56 days before randomisation

Exclusion Criteria:

* Diagnosis of any DSM-IV Axis I disorder other than those included in inclusion criteria above within 6 months before randomisation (e.g., alcohol dependence or psychoactive substance dependence not in full remission, concurrent organic mental disorder, or mental retardation [axis II diagnosis]) of a degree that may interfere with the patient's ability to co-operate.
* Previous stable use of high dosage of benzodiazepines during one year or more
* Significant neurological medical history (complicated head trauma as judged by the investigator, epilepsy, meningo-encephalitis)
* Use of the following medication:
* other antipsychotic drug than quetiapine within 28 days prior to randomisation
* a depot antipsychotic injection within two dosing intervals (for the depot) before randomisation (Visit 2)
* other psychoactive drugs within 14 days prior to randomisation (hypnotic or anxiolytic drugs, other than those allowed)
* Use of concomitant therapy likely to affect cognition, Medication prohibited 28 days prior to randomisation: benzodiazepines, amphetamines, reboxitin, atomoxinetine, buspiron, donepezil, duloxetine, galantamine, ginko biloba, memantine, methylphenidate, modafinil, rivastigmine, tacrine, smoking cessation therapy varencicline and any dosage form of nicotine replacement therapy. Medication prohibited 14 days prior to randomisation: irreversible monoamine oxidase inhibitors (MAOI), tricyclic antidepressants (TCA), biperiden, antoicholinergic agents (even if the indications are extra pyramidal symptoms or urinary symptoms)

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 75 (Actual)
Dates: Start 2010-11; Primary Completion 2011-08 (Actual); Study Completion 2011-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Eva Dencker Vansvik, Study Director — AstraZeneca
Locations (20):
- Research Site, Vienna, Austria
- Research Site, Middelfart, Denmark
- Germany (5):
  - Research Site, Berlin
  - Research Site, Bochum
  - Research Site, Hamburg
  - Research Site, München
  - Research Site, Rottweil
- Italy (11):
  - Research Site, Giarre, CT
  - Research Site, Genova, GE
  - Research Site, Lido di Camaiore, LU
  - Research Site, Barakaldo (vizcaya), Pais Vasco
  - Research Site, Tivoli, RM
  - Research Site, Sant'Arsenio, SA
  - Research Site, Sassari, SS
  - Research Site, Borgomanero
  - Research Site, Catania
  - Research Site, Roma
  - Research Site, Torre Annunziata
- Spain (2):
  - Research Site, Salamanca, Castille and León
  - Research Site, Zamora, Castille and León

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients were recruited at 20 study centres in 5 countries: Austria (1 site), Denmark (1 site), Germany (6 sites), Italy (9 sites) and Spain (3 sites). Recruitment started 2 November 2010 and was completed 29 June 2011. The last patient completed the study on 3 August 2011.
Pre-assignment Details: Screening (0 days to 14 days before enrolment), enrolment at Visit 1 (14 days to 3 days prior to randomisation), randomisation at Visit 2 after confirmation of eligibility. 75 patients were screened/enrolled. Of these, 9 were not randomised; 2 patients due to own decision to discontinue and 7 patients due to eligibility criteria not fulfilled.
Period: Period 1, First Intervention
Arm/Group | First Seroquel XR Then Seroquel IR | First Seroquel IR Then Seroquel XR
Started | 34 | 32
Completed | 31 | 29
Not Completed | 3 | 3
Not completed — Adverse Event | 2 | 1
Not completed — Protocol Violation | 0 | 1
Not completed — Withdrawal by Subject | 1 | 1
Period: Period 2, Second Intervention
Arm/Group | First Seroquel XR Then Seroquel IR | First Seroquel IR Then Seroquel XR
Started | 31 | 29
Completed | 31 | 29
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | First Seroquel XR Then Seroquel IR | First Seroquel IR Then Seroquel XR | Total
Number analyzed (Participants) | 34 | 32 | 66
Age Continuous [Number; unit: participants] — Of the 66 patients randomised to treatment with XR or IR only 65 patients took any study drug. One patient withdrew before taking any study drug. 65 patients were analysed for baseline age.
  participants
    between 18 and 29 years | 6 | 3 | 9
    Between 30 and 50 years | 26 | 28 | 54
    >50 years | 2 | 0 | 2
Age Continuous [Mean (Standard Deviation); unit: years] — Of the 66 patients randomised to treatment with XR or IR only 65 patients took any study drug. One patient withdrew before taking any study drug. 65 patients were analysed for baseline measure age.
  years | 38.6 (8.2) | 37.0 (5.2) | 37.8 (6.9)
Gender [Number; unit: participants] — Of the 66 patients randomised to treatment with XR or IR only 65 patients took any study drug. One patient withdrew before taking any study drug. 65 patients were analysed for baseline measure gender.
  participants
    Female | 11 | 9 | 20
    Male | 23 | 22 | 45
Region of Enrollment [Number; unit: participants]
  Spain | 1 | 1 | 2
  Denmark | 1 | 1 | 2
  Austria | 1 | 2 | 3
  Germany | 18 | 10 | 28
  Italy | 13 | 18 | 31

OUTCOME MEASURES:

1. Primary Outcome: Mean for Attentional Standardised Composite Score Based on Performance Scores From the CogState Test Battery Domains Detection (Speed of Processing)and Identification (Attention/Vigilance)
Description: Attentional standardised composite score: Standardised speed of performance score. Higher Score=better performance. Score range minus infinity to plus infinity. Measured at baseline (before study drug administration) and in Period 1 at 3 visits,(post 1),(post 2),(post 3), in a 5-day (maximum 8 day) period. (Last test day not earlier than after 10 days of randomised)and in Period 2 at 3 visits,(post 1),(post 2),(post 3), in a 5-day (maximum 8 day) period. Last test day not earlier than after 10 days of crossover treatment.
Time Frame: Period 1 at 3 visits,(post 1),(post 2),(post 3), in a 5-day (maximum 8 day) period. Period 2 at 3 visits,(post 1),(post 2),(post 3), in a 5-day (maximum 8 day) period.
Population: The per protocol set (PPS) is a subset of the FAS consisting of patients who fulfilled all inclusion criteria but none of the exclusion criteria, complied with study medication dosing scheme, did not violate any of the study restrictions and completed the study without protocol violation.
Measure: Mean (Standard Deviation); unit: standardised units
Groups:
- Seroquel XR; Seroquel IR: Patients that took Seroquel XR in arm XR-IR and arm IR-XR.
Arm/Group | Seroquel XR | Seroquel IR
Number analyzed (Participants) | 51 | 51
standardised units
  Post 1 | 0.002 (0.856) [-0.087 to 0.098] | -0.098 (0.983)
  Post 2 | -0.201 (1.054) | -0.131 (1.053)
  Post 3 | -0.194 (1.040) | -0.120 (1.100)

2. Secondary Outcome: Mean Treatment Satisfaction for Treatment Satisfaction Questionnaire of Medication (TSQM)
Description: TSQM is a 14-item questionnaire with 4 sub-scales: effectiveness of the medication; treatment side effects; convenience of the medication; global satisfaction with the medication. Scale range 0-100 for each sub-scale, higher=greater satisfaction/milder side effects/greater convenience/greater overall satisfaction.
  There are 2 measurement, (after the start of taking study drug) one at end of period 1 and one at end of period 2. That is one measurement per patient per treatment. The mean of all the patients is presented, one mean value per treatment group.
Time Frame: Before taking study drug, end of Period 1 and end of Period 2
Population: Full Analysis Set (FAS)used for efficacy analysis included all patients who in both study periods, received at least 1 dose of investigational product and for whom post-dose efficacy data was available.
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Seroquel IR: Patients that took Seroquel IR in arm XR-IR and arm IR-XR.
Arm/Group | Seroquel XR | Seroquel IR
Number analyzed (Participants) | 60 | 59
units on a scale
  Side Effects | 87.9 (20.5) | 81.5 (27.5)
  Effectiveness | 65.4 (16.8) | 62.2 (19.1)
  Convenience | 66.2 (19.3) | 63.6 (19.7)
  Overall Satisfaction | 63.0 (19.7) | 58.9 (21.1)

3. Secondary Outcome: Mean Daytime Cognitive Performance Using CogState: - Working Memory - Verbal Learning) -Reasoning and Problem Solving
Description: International Shopping List Task (ISLT): measures reasoning and problem solving. Min=minus infinity, max=plus infinity, higher score=better performance. Groton Maze Learning Test (GMLT): measures reasoning and problem solving. Min=minus infinity, max=plus infinity, lower score=better performance. Lower=better performance. One Back memory task (ONB: measures working memory, min=minus infinity, max=plus infinity, lower score=better performance.
Time Frame: as for outcome 1
Population: Per Protocol (PPS), subset of the FAS consisting of patients who fulfilled all of inclusion but none of exclusion criteria, complied with study medication dosing, did not violate any of the restrictions and completed the study without protocol violation.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Seroquel XR | Seroquel IR
Number analyzed (Participants) | 51 | 51
Units on a scale
  ISLT post 1 | 24.020 (5.746) [-0.220 to 1.055] | 23.588 (5.787)
  ISLT post 2 | 23.551 (4.899) [-2.714 to 3.791] | 23.152 (5.562)
  ISLT post 3 | 23.216 (5.360) [-0.026 to 0.009] | 22.920 (4.944)
  GMLT post 1 | 64.180 (29.822) | 61.040 (28.721)
  GMLT post 2 | 59.021 (21.257) | 56.956 (21.798)
  GMLT post 3 | 57.229 (24.162) | 57.300 (22.307)
  ONB post 1 | 2.875 (0.143) | 2.897 (0.134)
  ONB post 2 | 2.896 (0.151) | 2.896 (0.169)
  ONB post 3 | 2.894 (0.161) | 2.893 (0.154)

4. Secondary Outcome: Mean Overall Sedation as Measured by the Modified Bond-Lader Visual Analogue Scale (VAS) When Administered According to Label
Description: The modified Bond-Lader VAS: The degree of sedation was marked by the patient on a 100 mm VAS ranging between Alert (=0 mm) and Drowsy (=100 mm). The marked length in millimetres.
  There are 3 assessments made in each period (post 1, 2 and 3 for each period). That is three measurements per patient per treatment. The mean is an overall mean of all the recordings in all patients, one mean value per treatment group.
Time Frame: as for outcome 1
Population: The full analysis set (FAS) used for analysis of efficacy included all patients who, in both study periods, received at least one dose of investigational product and for whom post-dose efficacy data are available in both periods.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Seroquel XR | Seroquel IR
Number analyzed (Participants) | 60 | 60
units on a scale | 23.5 (19.0) | 28.6 (21.4)

5. Secondary Outcome: Mean Overall Sedation as Measured by the Stanford Sleepiness Scale When Administered According to Label
Description: Stanford Sleepiness Scale: The sleepiness was assessed by the patient on a 7 item rating scale ranging from 1 (Feeling active and vital) to 7 (Almost in reverie).
  There are 3 assessments made in each period (post 1, 2 and 3 for each period). That is three measurements per patient per treatment. The mean is an overall mean of all the recordings in all patients, one mean value per treatment group.
Time Frame: as for outcome 1
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Seroquel XR | Seroquel IR
Number analyzed (Participants) | 60 | 60
units on a scale | 2.4 (0.9) | 2.6 (1.0)

6. Secondary Outcome: Number of Dropouts.
Description: The number of patients who dropped out was counted.
Time Frame: Period 1 and Period 2
Population: The Safety analysis set was used, that is all patients who received at least one dose of study medication and for whom any post-dose safety data are available were included in the safety set.
Measure: Number; unit: participants
Groups:
- Seroquel XR: Patients treated with at least one dose of Seroquel XR
- Seroquel IR: Patients treated with at least one dose of Seroquel IR
Arm/Group | Seroquel XR | Seroquel IR
Number analyzed (Participants) | 34 | 31
participants
  Period 1 | 3 | 2
  Period 2 | 0 | 0

7. Secondary Outcome: Mean Ratio of Morning Plasma Concentration of Quetiapine and Nor-quetiapine for Quetiapine IR and Quetiapine XR, at Steady-state Conditions in the End of Each Treatment Period 1 and 2.
Description: The ratio was derived as individual plasma concentration of quetiapine divided by the plasma concentration of nor-quetiapine. The mean ratio was derived for each treatment, XR and IR, respectively.
Time Frame: End of Period 1, end of Period 2
Population: 21 patients for the FAS were analysed. This outcome measure was introduced as a protocol amendment after study start and plasma concentration was not measured in all patients. FAS is all patients who, in both study periods, received at least one dose of investigational product and for whom post-dose efficacy data are available in both periods.
Measure: Mean (Standard Deviation); unit: Ratio
Arm/Group | Seroquel XR | Seroquel IR
Number analyzed (Participants) | 21 | 21
Ratio | 1.941 (1.504) | 2.128 (2.369)

ADVERSE EVENTS:
Arm/Group | Seroquel XR | Seroquel IR
Serious Adverse Events (participants affected / at risk) | 0/63 | 0/62
Other Adverse Events (participants affected / at risk) | 4/63 | 4/62
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Seroquel XR (N=63) | Seroquel IR (N=62)
neutropenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
tachycardia (Cardiac disorders) | 0 (0) | 1 (1)
vertigo (Ear and labyrinth disorders) | 1 (1) | 0 (0)
fatigue (General disorders) | 0 (0) | 1 (1)
heart rate increase (Investigations) | 0 (0) | 1 (1)
dizziness (Nervous system disorders) | 0 (0) | 1 (1)
sedation (Nervous system disorders) | 1 (1) | 0 (0)
somnolence (Nervous system disorders) | 1 (1) | 2 (2)
delusion (Psychiatric disorders) | 0 (0) | 1 (1)
psychotic disorder (Psychiatric disorders) | 1 (1) | 0 (0)
sleep disorder (Psychiatric disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less